CLINICAL TRIAL: NCT00002325
Title: A Double-Blind, Placebo-Controlled Study of Fluconazole in the Prevention of Active Coccidioidomycosis and Other Systemic Fungal Infections in HIV-Infected Patients Living in the Coccidioidal Endemic Area
Brief Title: A Study of Fluconazole in the Prevention of Fungal Infections in HIV-Infected Patients Living in Areas Where Fungal Infections Are Common
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 012R; R-0266
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Mycoses; HIV Infections; Coccidioidomycosis
Keywords: Mycoses; Fluconazole; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Coccidioidomycosis
MeSH Terms: conditions — Mycoses; HIV Infections; Coccidioidomycosis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To compare the efficacy of fluconazole versus placebo in preventing the development of active coccidioidomycosis and other systemic fungal infections among HIV-infected patients with CD4 lymphocyte counts < 250 cells/mm3 who are living in the coccidioidal endemic area.

DETAILED DESCRIPTION:
Patients are randomized to receive either fluconazole or placebo daily.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 count < 250 cells/mm3.
* No active coccidioidomycosis or other fungal disease requiring systemic antifungal therapy.
* Residence in area considered to be endemic for Coccidioides immitis.
* Consent of parent or guardian if under legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Unable to take oral medication.
* Positive serum cryptococcal antigen.

Concurrent Medication:

Excluded:

* Systemic antifungal therapy.

Patients with the following prior conditions are excluded:

History of hypersensitivity to azole or imidazole compounds.

Prior Medication:

Excluded:

* Systemic antifungal agents within 2 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - McDowell Clinic, Phoenix, Arizona
  - Tucson Veterans Administration Med Ctr, Tucson, Arizona
  - Dr Lawrence Cone, Rancho Mirage, California